CLINICAL TRIAL: NCT00571701
Title: A Multicentered Randomized Study of Celebrex (Celecoxib) in Patients With Recurrent Respiratory Papillomatosis
Brief Title: Study of Celebrex (Celecoxib) in Patients With Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Iowa (Other); Eastern Virginia Medical School (Other); University of Alabama at Birmingham (Other); University of California, San Francisco (Other); Vanderbilt University (Other); Sanford Health (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1U01DC007946-01A2 (NIH); 1U01DC007946-01A2 (NIH); NCT00297999 (obsolete NCT alias)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: HPV; RRP
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- celecoxib first, then placebo (Active Comparator): Patients randomized to start celecoxib 6 months after enrollment. Then cross over to placebo after 1 year. Celecoxib dosing will be given orally 400mg once a day for adults, 200 mg once a day for pediatric patients between 12-25kg, 100mg once a day for pediatric patients < 12kg
  Interventions: Drug: celebrex (celecoxib); Drug: placebo
- Placebo first, then celecoxib (Placebo Comparator): Patients randomized to start placebo 6 months after enrollment. One placebo capsule will be taken orally once a day. Placebo will match appearance of active celecoxib capsules. Cross over to 12 months of treatment with celecoxib after 1 year.
  Interventions: Drug: celebrex (celecoxib); Drug: placebo

INTERVENTIONS:
Drug: celebrex (celecoxib) — Adults: 400 mg celebrex (celecoxib) daily Pediatrics: 100 mg celebrex (celecoxib) daily for weight between 12-25 kg or 200 mg Celebrex (celecoxib) daily for weight >25 kg
  Other Names: Celebrex
Drug: placebo — similar appearing capsules containing inert ingredients

SUMMARY:
This is a randomized double blind controlled study to determine if celebrex (celecoxib), a selective COX-2 inhibitor, can decrease the rate of recurrence in adult and pediatric patients with recurrent respiratory papillomatosis. All patients will be evaluated for disease severity at enrollment and at 3 month intervals for 30 months. After randomization, patients in the early treatment arm will begin celecoxib 6 months after enrollment. The delayed treatment arm will begin celecoxib 18 months after enrollment. All patients will receive celecoxib for 1 year. During the time that patients do not receive celecoxib, they will receive a placebo capsule with the same appearance. Follow-up visits will occur at three month intervals for the duration of the study.

DETAILED DESCRIPTION:
This is a randomized double blind placebo-controlled study,with plans to include 5 additional U.S. centers in the near future. The primary goal of this study is to determine whether celecoxib has efficacy in elimination or reduction of recurrent disease in patients with RRP. Our secondary goals are to determine whether continued celecoxib is required to maintain response, to correlate response with select patient demographics and with plasma levels of celecoxib. The study design encompasses a 30-month period, which can be divided into three segments:

Segment A: This is a 6 month run-in period in which all patients are assessed by direct laryngoscopy/bronchoscopy for disease severity, to permit growth rate stabilization and confirm accuracy of training of participating physicians. Patients will be treated by conventional surgery at three months and six months after enrollment.

Segment B: Patients begin 12 months of 400mg(adults), 100 mg (pediatric weight between 12 and 25 kg)or 200 mg (pediatric weight > 25kg) celecoxib daily or placebo treatment in addition to surgical removal of all papillomas at each 3 month interval. This segment directly tests the hypothesis that celecoxib is an efficacious treatment for moderate to severe RRP and forms the basis for the primary statistical analyses.

Segment C: The primary purpose of this segment is to determine whether gains made during celecoxib therapy are maintained after it is discontinued, or whether celecoxib will need to be taken indefinitely. This will be determined by a 12 month period on placebo after cessation of celecoxib for the early treatment group. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C. However, the placebo first group was given celecoxib so that they could gain any possible benefits equivalent to those that received the celecoxib first.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe disease, defined as:

Patients who have rapid regrowth of papillomas, requiring endoscopic removal at least 3 times within the past 12 months AND A papilloma growth rate from 0.03 to 0.06 (moderate) or >0.06 (severe) at time of initial direct endoscopy OR Having tracheal and/or bronchial or pulmonary papillomatosis (severe)

* Age > 2 years
* Gender- no restriction
* Race- no restriction

Exclusion Criteria:

* Fewer than 3 surgical procedures in previous year, without tracheal disease
* Age < 2 years
* Pregnancy, trying to become pregnant, breastfeeding or not willing to comply with birth control methods if sexually active female
* Serum creatinine > 1.5 X normal
* History of documented peptic ulcer disease or gastritis persisting despite treatment
* Abnormal liver function tests, as total bilirubin >1.5 X normal and SGOT > 3 X normal
* Allergy to NSAIDs, sulfa containing drugs or symptoms of Stevens-Johnson Syndrome
* Patients with connective tissue diseases such as SLE, Raynaud's or Systemic Sclerosis
* Patients with known diabetes
* Patients on warfarin, or on loop or thiazide diuretics
* Patients with a history of cardiovascular disease, myocardial infarct or stroke
* Patients with congestive heart failure
* Patients regularly taking > 81 mg of aspirin/day
* Patients with uncontrolled hypertension
* Patients with RRP associated malignancy currently receiving chemotherapy and/or radiation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettie M Steinberg, PhD, Principal Investigator — Long Island Jewish Medical Center
Locations (7):
- United States (7):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UCSF Medical Center, San Francisco, California
  - University of Iowa, Iowa City, Iowa
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Sanford Health /USD, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu R, Abramson AL, Shikowitz MJ, Dannenberg AJ, Steinberg BM. Epidermal growth factor-induced cyclooxygenase-2 expression is mediated through phosphatidylinositol-3 kinase, not mitogen-activated protein/extracellular signal-regulated kinase kinase, in recurrent respiratory papillomas. Clin Cancer Res. 2005 Sep 1;11(17):6155-61. doi: 10.1158/1078-0432.CCR-04-2664. PMID 16144915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 7 participating sites throughout the U.S. (locations in NY, VA, SD, AL, CA, IA and TN) that had investigators experienced in the treatment of this disease.
Pre-assignment Details: Patients initially entered a 6 month pre-treatment observation period prior to randomization into the 2 treatment arms. 9 subjects did not start the treatment period and are therefore not included in demographics or the results sections.
Groups:
- Celecoxib First (12 Months), Then Placebo (12 Months): Patients randomized to start celecoxib 6 months after enrollment. Then cross over to placebo after 1 year. Celecoxib dosing will be given orally 400mg once a day for adults, 200 mg once a day for pediatric patients between 12-25kg, 100mg once a day for pediatric patients < 12kg
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
- Placebo First (12 Months), Then Celecoxib (12 Months): Patients randomized to start placebo 6 months after enrollment. One placebo capsule will be taken orally once a day. Placebo will match appearance of active celecoxib capsules. Cross over to 12 months of treatment with celecoxib after 1 year.
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
Period: First Intervention 12 Months
Arm/Group | Celecoxib First (12 Months), Then Placebo (12 Months) | Placebo First (12 Months), Then Celecoxib (12 Months)
Started | 19 | 22
Completed | 16 | 21
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 1 | 0
Period: Second Intervention 12 Months
Arm/Group | Celecoxib First (12 Months), Then Placebo (12 Months) | Placebo First (12 Months), Then Celecoxib (12 Months)
Started | 16 | 21
Completed | 13 | 20
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib First, Then Placebo: Patients randomized to start celecoxib 6 months after enrollment. Then cross over to placebo after 1 year. Celecoxib dosing will be given orally 400mg once a day for adults, 200 mg once a day for pediatric patients between 12-25kg, 100mg once a day for pediatric patients < 12kg
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
- Placebo First, Then Celecoxib: Patients randomized to start placebo 6 months after enrollment. One placebo capsule will be taken orally once a day. Placebo will match appearance of active celecoxib capsules. Cross over to 12 months of treatment with celecoxib after 1 year.
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
- Total: Total of all reporting groups
Arm/Group | Celecoxib First, Then Placebo | Placebo First, Then Celecoxib | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Customized [Number; unit: participants]
  Age < 20 | 9 | 11 | 20
  Age 20 - < 40 | 3 | 9 | 12
  Age 40 and above | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 19 | 36
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Papilloma Growth Rate at 12 Month Measurement Compared to Baseline
Description: Change in mean growth rates during the last 3 months of the first treatment period compared to the mean values at baseline. Endoscopy and removal of all tumor was done every 3 months. Growth rate is calculated as the scored amount of papilloma recurrence in a 3 month period divided by the exact number of days since last endoscopy and removal of all tumor.
Time Frame: Baseline to 12 months
Population: All patients in each arm who completed the first 1 year treatment period. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Mean (Standard Deviation); unit: percent change in mean growth rate
Groups:
- Celecoxib First, Then Placebo: Patients randomized to start celecoxib. Then cross over to placebo after 1 year. Celecoxib dosing will be given orally 400mg once a day for adults, 200 mg once a day for pediatric patients between 12-25kg, 100mg once a day for pediatric patients < 12kg
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
- Placebo First, Then Celecoxib: Patients randomized to start placebo. One placebo capsule will be taken orally once a day. Placebo will match appearance of active celecoxib capsules. Cross over to 12 months of treatment with celecoxib after 1 year.
  celebrex (celecoxib): Adults: 400 mg daily Pediatrics: 100 mg daily for weight between 12-25 kg or 200 mg daily for weight >25 kg
Arm/Group | Celecoxib First, Then Placebo | Placebo First, Then Celecoxib
Number analyzed (Participants) | 16 | 21
percent change in mean growth rate | -5.4 (50.0) | -15.2 (67.3)
Statistical Analysis 1: Comparison: Celecoxib First, Then Placebo vs Placebo First, Then Celecoxib; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent of Patients With Positive Response to Treatment
Description: Percent of patients with reduction in papilloma growth rate greater than 50% during the last 3 months of first treatment period compared to baseline
Time Frame: Baseline to 12 months
Population: All patients that completed first treatment period. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Number; unit: percent responders
Arm/Group | Celecoxib First (12 Months), Then Placebo (12 Months) | Placebo First (12 Months), Then Celecoxib (12 Months)
Number analyzed (Participants) | 16 | 21
percent responders | 12.5 | 28.6
Statistical Analysis 1: Comparison: Celecoxib First (12 Months), Then Placebo (12 Months) vs Placebo First (12 Months), Then Celecoxib (12 Months); Test type: Superiority or Other; p = 0.43, Fisher Exact

3. Secondary Outcome: Effect of Gender on Percent of Patients With Reduction in Papilloma Growth Rate Greater Than 50%.
Description: Percent of patients of each gender with reduction in papilloma growth rate greater than 50% during the last 3 months of first treatment period compared to baseline
Time Frame: Baseline to12 months
Population: All patients who completed first treatment period. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Number; unit: percent responders
Groups:
- Celecoxib First - Males: Males treated with celecoxib during the first treatment period
- Placebo First- Males: Males treated with placebo during the first treatment period
- Celecoxib First- Females: Females treated with celecoxib during the first treatment period
- Placebo First- Females: Females treated with placebo during the first treatment period
Arm/Group | Celecoxib First - Males | Placebo First- Males | Celecoxib First- Females | Placebo First- Females
Number analyzed (Participants) | 8 | 15 | 8 | 6
percent responders | 12.50 | 40.00 | 12.50 | 0.00
Statistical Analysis 1: Comparison: Celecoxib First - Males vs Placebo First- Males vs Celecoxib First- Females vs Placebo First- Females; Test type: Superiority or Other; p > 0.3, Fisher Exact — Adjusted for multiple comparisons

4. Secondary Outcome: Effect of Juvenile Versus Adult Disease Onset on Percent of Patients With Reduction in Papilloma Growth Rate Greater Than 50%.
Description: Percent of juvenile versus adult onset patients with reduction in papilloma growth rate greater than 50% during the last 3 months of first treatment period compared to baseline.
Time Frame: Baseline to 12 months
Population: Analysis conducted on all patients who completed first treatment period. Juvenile onset is defined as <18 years of age at time of diagnosis. Age of disease onset for 2 patients was not available. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Number; unit: percentage of responders
Groups:
- Celecoxib First- Juvenile Onset: Juvenile-onset subjects treated with celecoxib during the first treatment period
- Placebo First- Juvenile-onsent: Juvenile-onset subjects treated with placebo during first treatment period
- Celecoxib First - Adult Onset: Adult-onset subjects treated with celecoxib during the first treatment period
- Placebo First- Adult-onset: Adult-onset subjects treated with placebo during the first treatment
Arm/Group | Celecoxib First- Juvenile Onset | Placebo First- Juvenile-onsent | Celecoxib First - Adult Onset | Placebo First- Adult-onset
Number analyzed (Participants) | 8 | 13 | 8 | 6
percentage of responders | 12.50 | 7.69 | 12.50 | 33.33
Statistical Analysis 1: Comparison: Celecoxib First- Juvenile Onset vs Placebo First- Juvenile-onsent vs Celecoxib First - Adult Onset vs Placebo First- Adult-onset; Test type: Superiority or Other; p = 1.00, Fisher Exact — Adjusted for multiple comparisons

5. Secondary Outcome: Effect of HPV 6 Versus HPV 11 on Percent of Patients With Reduction in Papilloma Growth Rate Greater Than 50%
Description: Percent of patients with HPV 6 versus patients with HPV 11 with reduction in papilloma growth rate greater than 50% during the last 3 months of first treatment period compared to baseline.
Time Frame: Baseline to 12 months
Population: Analysis conducted on all patients with HPV 6 or 11 infection who completed first treatment period. One patient with both HPV 6 and 11 and one patient with neither 6 or 11 were excluded. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Number; unit: percent of responders
Groups:
- Celecoxib First - HPV 6: Subjects infected with HPV 6 treated with celecoxib during the first treatment period
- Placebo First- HPV 6: Subjects infected with HPV 6 treated with placebo during first treatment period
- Celecoxib First- HPV 11: Subjects infected with HPV 11 treated with celecoxib during the first treatment period
- Placebo First- HPV 11: Subjects infected with HPV 11 treated with placebo during the first treatment period
Arm/Group | Celecoxib First - HPV 6 | Placebo First- HPV 6 | Celecoxib First- HPV 11 | Placebo First- HPV 11
Number analyzed (Participants) | 11 | 14 | 4 | 5
percent of responders | 9.09 | 42.86 | 25.00 | 0.00
Statistical Analysis 1: Comparison: Celecoxib First - HPV 6 vs Placebo First- HPV 6 vs Celecoxib First- HPV 11 vs Placebo First- HPV 11; Test type: Superiority or Other; p > 0.5, Fisher Exact — Adjusted for multiple comparisons

6. Secondary Outcome: Correlation Between Mean Plasma Level of Celecoxib and Response.
Description: Mean plasma levels of celecoxib over months 3-12 in first treatment period correlated with reduction in papilloma growth rate greater than 50% during the last 3 months of first treatment period compared to baseline.
Time Frame: Baseline to 12 months
Population: All patients who were randomized to receive celecoxib first and completed the first treatment period. This is not a traditional cross-over study because we expected a sustained effect therefore no efficacy studies were done in segment C.
Measure: Mean (Full Range); unit: pg. celecoxib/ml. plasma
Groups:
- Responders: Subjects randomized to celecoxib first with response greater than 50% at end of first treatment period relative to mean disease severity prior to treatment.
- Non-responders: Subjects randomized to celecoxib first with response less than 50% at end of first treatment period relative to mean disease severity prior to treatment.
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 2 | 14
pg. celecoxib/ml. plasma | 151.3 [126.6 to 176.00] | 543.41 [10.00 to 2422.50]
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p > 0.56, t-test, 2 sided

7. Secondary Outcome: Maintenance of Response Following Discontinuation of Celecoxib
Description: Percent of patients who responded to celecoxib with increase in papilloma growth rate of no greater than 0.01 at end of second treatment period compared to growth rate at end of first treatment period.
Time Frame: End of first treatment period (month 12) to end of second treatment period (month 24)
Population: All patients with complete response to celecoxib in first treatment period who completed the second treatment period where they received placebo. Because the number of responders was so small, no statistical analysis was performed.
Measure: Number; unit: percent of patients
Groups:
- Celecoxib Responders-maintained: Subjects randomized to celecoxib first with response greater than 50% at end of first treatment period that maintained response at end of second treatment.
- Celecoxib Responders- Not Maintained: Subjects randomized to celecoxib first with response greater than 50% at end of first treatment period whose papilloma growth rate worsened by more than 0.01 at end of second treatment period.
Arm/Group | Celecoxib Responders-maintained | Celecoxib Responders- Not Maintained
Number analyzed (Participants) | 2 | 0
percent of patients | 100 |

ADVERSE EVENTS:
Time Frame: AE reporting included all subjects who received at least three doses of study intervention. AE reporting was done throughout the entire 2 year period after randomization and also included up to approximately 30 days after the last dose of study drug was taken.
Groups:
- Celecoxib: Patients who received celecoxib for 12 months during either time period
- Placebo: Patients who received placebo for 12 months during either time period
Arm/Group | Celecoxib | Placebo
Serious Adverse Events (participants affected / at risk) | 3/40 | 2/39
Other Adverse Events (participants affected / at risk) | 16/40 | 18/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=40) | Placebo (N=39)
death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient withdrew during 1st study period, died of pulmonary pneumonia secondary to RRP associated lung cancer 3 months after her last dose of study drug
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — pneumonia resulting in inpatient hospitalization, 2 subjects had known pulmonary RRP and third patient had a tracheotomy
palpable lymph node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Patient with long-history of pulmonary RRP found to have palpable lymph node- needle biopsy revealed atypical findings and additional findings confirmed metastatic RRP associated lung cancer
influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Resulted in inpatient hospitalization for this patient due to dehydration secondary to diarrhea and vomiting as a result of the influenza
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=40) | Placebo (N=39)
abdominal pain (Gastrointestinal disorders) | 4 | 5 — Includes AEs reported as abdominal discomfort, abdominal pain, abdominal pain upper, dyspepsia, flatulence, gastritis and stomach infection
nausea or vomiting (Gastrointestinal disorders) | 2 | 5
non-cardiac chest discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 4 — AE term includes cough, chest discomfort
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 | 9 — AE terms include increased nasal secretions, rhinitis, strep infection, croup and sinusitis
pyrexia (General disorders) | 2 | 5 — elevated temperature
diarrhea (Gastrointestinal disorders) | 4 | 3

LIMITATIONS AND CAVEATS:
Rare prevalence of moderate to severe recurrent respiratory papillomatosis (estimated at 1:1million) limited enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No